CLINICAL TRIAL: NCT03604809
Title: Guided Occupational Therapist Cognitive Interventions in Critically Ill Patients
Acronym: GOTCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alberta Health Services, Calgary (Other)
Responsible Party: Principal Investigator, Kirsten Deemer, NP, Critical Care Nurse Practitioner, Alberta Health Services, Calgary
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2018-06-18; First posted 2018-07-30 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: All investigators, with the exception of the occupational therapist, will be blinded to participant randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OT Guided Cognitive Interventions (Experimental): Occupational Therapy interventions will be adjusted according to the patient's Richmond Agitation and Sedation Scale (RASS).
  Interventions: Other: OT Guided Cognitive Interventions
- Usual Care (No Intervention): This will be the standard of care currently provided for delirium prevention within the Department of Critical Care Medicine in Calgary using the ABCDEF bundled approach.

INTERVENTIONS:
Other: OT Guided Cognitive Interventions — RASS is defined as the level of sedation and agitation of a patient. Cognitive interventions are evidence based strategies that enhance the cognition of patients and include memory training using visual imagery; metacognitive training using self-awareness and self-regulation approaches for recovery of executive functioning; and neuropsychological rehabilitation to help improve cognitive and functional deficits. Interventions will be adjusted according to the RASS score. Cognitive interventions include discussion of patient status and education of family around reorientation, cognitive screening and graded exercises according to patient ability. The deepest levels of sedation and highest levels of agitation will be included in the intervention arm.
  Interventions will be provided by the Occupational Therapist; Monday to Friday, BID, 20 minutes per session, for the duration of ICU admission.
  Arms: OT Guided Cognitive Interventions

SUMMARY:
Title: Guided Occupational Therapist (OT) Cognitive Interventions for Critically Ill Patients

Short Title: GOTCI

Methodology: Randomized Control Trial

Study Duration: 12-15 months

Study Centre: Single Center - South Health Campus, ICU, Calgary, Alberta, Canada

Objectives: The aim for this study is to evaluate the effect of specific OT guided cognitive interventions on delirium in adult critically ill patients.

Number of Subjects: 112

Primary Outcome: Delirium Prevalence and Duration

Secondary Outcomes: Cognitive function, physical function, quality of life, ICU length of stay, hospital length of stay and days of mechanical ventilation.

Inclusion Criteria: Adult Critically Ill Patients admitted to South Health Campus ICU, Calgary, Alberta

Type of Intervention: OT guided cognitive intervention based on RASS score

Dose: One on one therapeutic sessions with an OT. Five days a week, Monday to Friday, between 0800-1600. There will be twice daily sessions for 20 minutes each.

Duration of administration: Cognitive Therapy to be initiated Monday to Friday, for the duration of participant ICU admission.

Reference therapy: Standard of care within the Department of Critical Care Medicine in Calgary is delirium prevention strategies using the ABCDEF bundled approach.

Statistical Methodology: Descriptive statistics (mean, median, proportion) will be employed to describe the study population. The primary outcome of delirium prevalence will be explored using multivariable logistic regression, which will provide an estimate of the odds ratio and accompanying 95% confidence intervals. Both per protocol and intent to treat analyses will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Adult medical/surgical critically ill patients admitted to the South Health Campus ICU in Calgary, Alberta during designated 6-month study period.

Exclusion criteria as follows:

1. Primary Direct Brain Injury
2. Prior diagnosis of dementia-related illness
3. Prior diagnosis of developmental disability
4. Pre-existing cognitive impairment
5. Requiring palliative care
6. In ICU for less than 48 hours
7. Non-English speaking
8. Severe communication disorders
9. Non-critically ill Plasma Exchange Therapy patients
10. Severe hearing or visual impairment
11. ICU to ICU transfers
12. COVID-19 positive patients

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Delirium Prevalence and Duration | From date of patient enrolment to ICU discharge, an average of 6.7 days.
  Ever Delirium: Measured using the Intensive Care Delirium Screening Checklist (ICDSC). If the patient has a positive score in the ICDSC at any point during the patient's ICU stay then the patient is considered to have delirium and qualifies for Ever Delirium.
  Delirium Duration: Number of days the patient has a positive score on the ICDSC. This does not have to be consecutive days.

SECONDARY OUTCOMES:
Cognitive Function | Measured within 24 hours of patient ICU admission and again after the treatment period is completed which is an average of 6.7 days.
  Johns Hopkins Adapted Cognitive Exam (ACE)
  o The Adapted Cognitive Exam is the first valid and reliable examination for the assessment and quantification of cognition in critically ill patients. It provides a useful, objective tool that can be used by any member of the interdisciplinary critical care team to support clinical assessment and research efforts.
ICU length of stay | ICU admission date to ICU discharge date is the time the patient will be given the treatment which is an average of 6.7 days.
  Dates will be obtained from electronic medical charts. I.e. Sunrise Clinical Manager.
Physical Function | Measured within 48 hours of ICU admission and again after the treatment period is completed which is an average of 6.7 days.
  The Functional Status Score for the ICU (FSS-ICU). The Functional Status Score for the ICU (FSS-ICU) is an assessment of physical function specifically designed for ICU patients. It is scored based on 5 mobility domains (rolling in bed, lying to sitting, sitting balance, sitting to standing and walking) and the level of assistance the patient requires to complete the task. Each item is out of 7, with total scores ranging from 0-35 and a high score correlating to high function. The FSS-ICU has good validity when compared to other functional measures in the ICU, it has been demonstrated to have good interrater reliability and has minimal floor and ceiling effect.
Quality of Life using the EQ5D-5L (EuroQual 5 Dimensions-5 Levels). This is a health quality of life measure assessing five domains; mobility, self-care, usual activities, pain/discomfort and anxiety/depression. | Measured after the treatment period is completed (within 24 hours of discharge) which is an average of 6.7 days.
  The 5 Level EQ 5D version is a standardized measure of health status developed by the EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal (Van Reenan & Janssen, 2015). It covers five dimensions; mobility, self-care, usual activities, pain/discomfort and anxiety/depression which are measured with one of five response options (no problems, slight problems, moderate problems, severe problems, and extreme problems). A total of 3125 possible health states is defined in this way. Each state is referred to in terms of a 5 digit code. For example, state 11111 indicates no problems on any of the 5 dimensions, while state 12345 indicates no problems with mobility, slight problems with washing or dressing, moderate problems with doing usual activities, severe pain or discomfort and extreme anxiety or depression (Reenan & Janssen, 2015, p. 9). The EQ5D-5L also includes a visual analog scale to measure health state (0-100).
Days of Mechanical Ventilation | Measured on day 1 of mechanical ventilation through to day of extubation (cessation of mechanical ventilation), an average of 4 days.
  Dates will be obtained from electronic medical charts. i.e. Metavision
Length of Hospital Stay | Up to 6 months
  Date of hospital admission and discharge will be obtained from electronic medical chart. i.e. Sunrise Clinical Manager.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Oviatt, MScPT PT, Principal Investigator — Alberta Health services; Michelle Parsons, BHScPT PT, Principal Investigator — Alberta Health services; Kirsten Fiest, PhD, Principal Investigator — University of Calgary, Alberta Health Services; Karolina Herold, MN RN, Principal Investigator — Alberta Health services; Juan Posadas, MD, Principal Investigator — University of Calgary, Alberta Health Services; Brittany Myhre, MScOT OT, Principal Investigator — Alberta Health services; Andrea Soo, PhD, Principal Investigator — University of Calgary
Locations (1):
- South Health Campus Intensive Care Unit, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lewin JJ 3rd, LeDroux SN, Shermock KM, Thompson CB, Goodwin HE, Mirski EA, Gill RS, Mirski MA. Validity and reliability of The Johns Hopkins Adapted Cognitive Exam for critically ill patients. Crit Care Med. 2012 Jan;40(1):139-44. doi: 10.1097/CCM.0b013e31822ef9fc. PMID 21926576
- [Background] Huang M, Chan KS, Zanni JM, Parry SM, Neto SG, Neto JA, da Silva VZ, Kho ME, Needham DM. Functional Status Score for the ICU: An International Clinimetric Analysis of Validity, Responsiveness, and Minimal Important Difference. Crit Care Med. 2016 Dec;44(12):e1155-e1164. doi: 10.1097/CCM.0000000000001949. PMID 27488220
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Bergeron N, Dubois MJ, Dumont M, Dial S, Skrobik Y. Intensive Care Delirium Screening Checklist: evaluation of a new screening tool. Intensive Care Med. 2001 May;27(5):859-64. doi: 10.1007/s001340100909. PMID 11430542
- [Background] van den Boogaard M, Schoonhoven L, Maseda E, Plowright C, Jones C, Luetz A, Sackey PV, Jorens PG, Aitken LM, van Haren FM, Donders R, van der Hoeven JG, Pickkers P. Recalibration of the delirium prediction model for ICU patients (PRE-DELIRIC): a multinational observational study. Intensive Care Med. 2014 Mar;40(3):361-9. doi: 10.1007/s00134-013-3202-7. Epub 2014 Jan 18. PMID 24441670
- [Background] Wassenaar A, Rood P, Boelen D, Schoonhoven L, Pickkers P, van den Boogaard M. Feasibility of Cognitive Training in Critically Ill Patients: A Pilot Study. Am J Crit Care. 2018 Mar;27(2):124-135. doi: 10.4037/ajcc2018467. PMID 29496769
- [Background] Deemer K, Zjadewicz K, Fiest K, Oviatt S, Parsons M, Myhre B, Posadas-Calleja J. Effect of early cognitive interventions on delirium in critically ill patients: a systematic review. Can J Anaesth. 2020 Aug;67(8):1016-1034. doi: 10.1007/s12630-020-01670-z. Epub 2020 Apr 24. PMID 32333291
- [Derived] Deemer K, Myhre B, Oviatt S, Parsons M, Watson M, Zjadewicz K, Soo A, Fiest K, Posadas-Calleja J. Occupational therapist-guided cognitive interventions in critically ill patients: a feasibility randomized controlled trial. Can J Anaesth. 2023 Jan;70(1):139-150. doi: 10.1007/s12630-022-02351-9. Epub 2022 Nov 16. PMID 36385466